CLINICAL TRIAL: NCT01237054
Title: A Pilot Study of Novel Imaging Modalities in Monoclonal Gammopathy of Undetermined Significance (MGUS), Smoldering Multiple Myeloma (SMM), and Multiple Myeloma (MM)
Brief Title: Imaging in MGUS, SMM and MM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter Choyke, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 110020; 11-C-0020
Record Dates: First submitted 2010-11-06; First posted 2010-11-09 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance
Keywords: 18-FDG PET/CT; Abnormal Plasma Cells; Serum Free Light-Chain Abnormality; Serum M-Protein; DCE-MRI; Multiple Myeloma; Smoldering Multiple Myeloma; SMM; MM
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imaging in MGUS, SMM, and MM (Experimental): Participants will have three imaging studies on separate days: a standard positron emission tomography/computed tomography scan (18-FDG PET/CT), a PET/CT scan with an experimental sodium fluoride-based drug (18-NaF PET/CT), and magnetic resonance imaging (DCE-MRI).
  Interventions: Drug: 18-NaF PET; Other: DCE-MRI; Drug: 18-FDG PET/CT

INTERVENTIONS:
Drug: 18-NaF PET — The patient will receive 5mCi of F-18 NaF IV (intravenous) bolus, followed by a ~20 ml saline (sodium chloride IV infusion 0.9% w/v) flush over a period of ~20 seconds. Serial dynamic imaging (2 minutes/bed position) will be obtained over a 1-hour period. The patient will be permitted an imaging break until a static PET/CT is performed beginning at 2-hours post F-18 NaF injection.
Other: DCE-MRI — An FDA (Food and Drug Administration) approved gadolinium chelate (e.g. Magnevist, Berlex Laboratories, NJ, USA) will be administered intravenously at 3 cc/sec using an automated pump injector (Medrad, Pittsburgh, PA, USA).
Drug: 18-FDG PET/CT — The 18F-FDG injection procedure will be injected and be followed by a ~20 ml saline (sodium chloride IV infusion 0.9% w/v) flush over a period of ~20 seconds. The injection site will be evaluated pre- and post administration for any reaction (e.g. bleeding, hematoma, redness, or infection). Whole body (vertex to toes) static PET/CT imaging will be performed beginning at 1-hour, and again at 2-hours post injection.

SUMMARY:
Background:

- Recent studies have shown that the premalignant conditions monoclonal gammopathy of undetermined significance (MGUS) and smoldering multiple myeloma (SMM) have a high risk of progressing to multiple myeloma (MM). There are currently no known effective treatments to prevent MGUS or SMM from developing into MM, and there are no known tests for determining whether an individual with MGUS or SMM will develop MM. Researchers are investigating new and improved imaging techniques that may be able to better detect the progression of MGUS or SMM into MM.

Objectives:

* To compare the results of three imaging techniques in individuals with MGUS, SMM, and MM.
* To correlate the information from the imaging studies with established clinical markers of progression from MGUS/SMM to MM.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with monoclonal gammopathy of undetermined significance, smoldering multiple myeloma, or multiple myeloma.

Design:

* Participants will be screened with a physical examination and medical history, and will provide baseline blood, urine, and bone marrow samples before beginning the imaging studies.
* Participants will have three imaging studies on separate days: a standard 18-fludeoxyglucose positron emission tomography/computed tomography scan (18-FDG PET/CT), a PET/CT scan with an experimental sodium fluoride-based drug (18-NaF PET/CT), and dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI).
* Participants will be closely monitored during each scan, and will provide additional blood samples before and after the scans.
* Participants may provide additional blood, urine, tissue, and bone marrow samples for optional research studies.

DETAILED DESCRIPTION:
Background:

* Multiple myeloma (MM) is a plasma cell neoplasm with a median survival of 3-4 years.
* Monoclonal gammopathy of undetermined significance (MGUS) and smoldering myeloma (SMM) are premalignant plasma cell proliferative disorders characterized by elevated monoclonal protein and bone marrow plasma cells. MGUS affects 3.2% of Caucasians over the age of 50 and has a 1% annual risk of progression to MM.

Approximately 3000 cases of SMM are diagnosed annually with a 10% annual risk of progression to MM.

* Currently, it is not possible to predict which patients will progress to MM.
* Novel imaging modalities (FDG-PET, 18-NaF PET and DCE-MRI) may improve our ability to predict patients who are at high risk of progression.

Objectives:

* To compare the results of imaging modalities (18-NaF PET/CT, 18-FDG PET/CT, and DCE-MRI) in patients with MGUS, SMM, and MM.
* To correlate the imaging studies with established clinical markers of progression from MGUS/SMM to MM, including serum M-protein, percentage of plasma cells in the bone marrow, serum free light-chain abnormalities and immunoparesis, and ratio of normal/abnormal plasma cells in the bone marrow by flow cytometry.

Eligibility:

* A confirmed diagnosis of MGUS, SMM or MM (based on IMWG (International Myeloma Working Group) diagnostic criteria)
* Age greater than or equal to 18 years
* ECOG (Eastern Cooperative Oncology Group) performance status in the range of 0-2

Design:

* This is a cross-sectional pilot study of patients with MGUS, SMM or MM.
* Following initial evaluation and confirmation of diagnosis, baseline studies including skeletal survey will be done.
* Subsequently 18-NaF PET/CT, 18-FDG PET/CT and DCE-MRI imaging will be done in all the patients.
* 10 MGUS, 11 SMM and 10 MM patients will be enrolled on this protocol.
* Patients may donate cellular products or tissues as appropriate for research purposes.
* Almost all MGUS and SMM patients will be followed clinically as part of 10-C-0096:

Natural History Study of Monoclonal Gammopathy of Undetermined Significance (MGUS) and Smoldering Myeloma (SMM).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of MGUS, SMM and MM will be made in accordance with the clinical diagnostic criteria set forth by the International Myeloma Working Group.2. The diagnoses will be confirmed by laboratory tests, serum/urine protein electrophoresis, immunofixation and light-chain assays, a skeletal survey, or immunohistochemistry analyses of the bone marrow biopsy, or a combination of these.
* Age greater than or equal to 18 years.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-2.
* The patient must be competent to sign an informed consent form.
* Creatinine less than 2.5 ULN or eGFR (estimated glomerular filtration rate) greater than 30

EXCLUSION CRITERIA:

* A medical history of other malignancy (apart from basal cell carcinoma of the skin or in situ cervical carcinoma; also, for MM patients this does not include MM) except if the patient has been free of symptoms and without active therapy during at least the previous 5 years.
* Female subject is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-10-17 (Actual); Primary Completion 2011-08-09 (Actual); Study Completion 2011-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Choyke, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] International Myeloma Working Group. Criteria for the classification of monoclonal gammopathies, multiple myeloma and related disorders: a report of the International Myeloma Working Group. Br J Haematol. 2003 Jun;121(5):749-57. PMID 12780789
- [Background] Kristinsson SY, Landgren O, Dickman PW, Derolf AR, Bjorkholm M. Patterns of survival in multiple myeloma: a population-based study of patients diagnosed in Sweden from 1973 to 2003. J Clin Oncol. 2007 May 20;25(15):1993-9. doi: 10.1200/JCO.2006.09.0100. Epub 2007 Apr 9. PMID 17420512
- [Background] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015
- [Derived] Bhutani M, Turkbey B, Tan E, Korde N, Kwok M, Manasanch EE, Tageja N, Mailankody S, Roschewski M, Mulquin M, Carpenter A, Lamping E, Minter AR, Weiss BM, Mena E, Lindenberg L, Calvo KR, Maric I, Usmani SZ, Choyke PL, Kurdziel K, Landgren O. Bone marrow abnormalities and early bone lesions in multiple myeloma and its precursor disease: a prospective study using functional and morphologic imaging. Leuk Lymphoma. 2016 May;57(5):1114-21. doi: 10.3109/10428194.2015.1090572. Epub 2016 Apr 7. PMID 26690712
- [Derived] Bhutani M, Turkbey B, Tan E, Kemp TJ, Pinto LA, Berg AR, Korde N, Minter AR, Weiss BM, Mena E, Lindenberg L, Aras O, Purdue MP, Hofmann JN, Steinberg SM, Calvo KR, Choyke PL, Maric I, Kurdziel K, Landgren O. Bone marrow angiogenesis in myeloma and its precursor disease: a prospective clinical trial. Leukemia. 2014 Feb;28(2):413-6. doi: 10.1038/leu.2013.268. Epub 2013 Sep 18. No abstract available. PMID 24045500

RESULTS

PARTICIPANT FLOW:
Groups:
- Imaging in MGUS, SMM, and MM: Participants will have three imaging studies on separate days: a standard positron emission tomography/computed tomography scan (18-FDG PET/CT), a PET/CT scan with an experimental sodium fluoride-based drug (18-NaF PET/CT), and magnetic resonance imaging (DCE-MRI).
  18-NaF PET: The patient will patient will receive 5mCi of F-18 NaF IV bolus, followed by a ~20 ml saline (sodium chloride IV infusion 0.9% w/v) flush over a period of ~20 seconds. Serial dynamic imaging (2 minutes/bed position) will be obtained over a 1-hour period. The patient will be permitted an imaging break until a static PET/CT is performed beginning at 2-hours post F-18 NaF injection. DCE-MRI: An FDA approved gadolinium chelate (e.g. Magnevist, Berlex Laboratories, NJ, USA) will be administered intravenously at 3 cc/sec using an automated pump injector (Medrad, Pittsburgh, PA, USA).18-FDG PET/CT: The 18F-FDG injection procedure will be injected and be followed by a ~20 ml saline flush over a period of ~20 sec.
Period: Overall Study
Arm/Group | Imaging in MGUS, SMM, and MM
Started | 31
Completed | 30
Not Completed | 1
Not completed — imaging 10C0096 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imaging in MGUS, SMM, and MM
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.89 (10.58)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Positive and Negative 18F-FDG PET CT and F18-NaF PET CT Imaging Results in Individuals With MGUS, SMM, and MM.
Description: 18F-FDG PET CT and F18-NaF PET CT imaging results were compared in participants with MGUS, SMM, and MM. Lesions were considered positive if focal uptake corresponded to lesions identified on CT for NaF and negative if no uptake seen in lesions. Criteria to define FDG positivity included parameters published by Zamagni et al with focal abnormal uptake more intense than background.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Groups:
- MGUS (Monoclonal Gammopathy of Undetermined Significance): MGUS (Monoclonal gammopathy of undetermined significance) is a premalignant plasma cell proliferative disorder.
- SMM (Smoldering Multiple Myeloma): Smoldering multiple myeloma (SMM)is a premalignant plasma cell proliferative disorder.
- MM (Multiple Myeloma): Multiple myeloma is a plasma cell neoplasm.
Arm/Group | MGUS (Monoclonal Gammopathy of Undetermined Significance) | SMM (Smoldering Multiple Myeloma) | MM (Multiple Myeloma)
Number analyzed (Participants) | 10 | 10 | 10
Participants
  Positive 18F-FDG PET CT result | 0 | 1 | 5
  Negative 18F-FDG PET CT result | 10 | 9 | 5
  Positive F18-NaF PET CT result | 0 | 0 | 9
  Negative F18-NaF PET CT result | 10 | 10 | 1

2. Primary Outcome: Count of Participants With Positive DCE-MRI Imaging Results
Description: DCE-MRI, an FDA approved gadolinium chelate (e.g. Magnevist, Berlex Laboratories, NJ, USA) will be administered intravenously at 3 cc/sec using an automated pump injector (Medrad, Pittsburgh, PA, USA). The criteria was presence of early and diffuse hyper-enhancement compared to the surrounding bone marrow. The pattern of marrow involvement on MRI was characterized as: (1) normal when there was no evidence of abnormal signal intensity; (2) focal, which consisted of localized areas of abnormal marrow; the lesions are darker than yellow marrow and slightly darker than or isointense to red marrow on T1-weights images; (3) diffuse, in which normal bone marrow signal intensity is completely absent, the intervertebral disks appear brighter than or isointense to the diseased marrow; and finally (4) heterogeneous that consists of innumerable small foci of disease on a background of intact marrow, with small dark lesions on T1-weighted images, which become bright on T2-weighted image.
Time Frame: 60 days
Population: Missing means the imaging test was not done. Unclear means it is indeterminate whether an imaging result is positive or negative.
Measure: Count of Participants; unit: Participants
Arm/Group | MGUS (Monoclonal Gammopathy of Undetermined Significance) | SMM (Smoldering Multiple Myeloma) | MM (Multiple Myeloma)
Number analyzed (Participants) | 10 | 10 | 10
Participants
  Positive | 1 | 1 | 9
  Negative | 9 | 9 | 0
  Missing | 0 | 0 | 1
  Unclear | 0 | 0 | 0

3. Secondary Outcome: Comparison of Serum Angiogenic Markers Ang2 (Angiopoietin), G-CSF (Granulocyte-colony Stimulating Factor), Follistatin, HGF (Hepatocyte Growth Factor), FGF-1, Endothelin 1, and VEGF-A (Vascular Endothelial Growth Factor-A) Between MGUS and SMM/MM Groups
Description: The assay was performed according to the manufacture's protocol, and all samples were diluted 1:3. Cytokine values were calculated using a five-parameter standard curve with Bio-Plex Manager 6.1.
Time Frame: 60 days
Population: Serum was not available for three patients in the SMM group.
Measure: Mean (Standard Error); unit: pg/ml
Groups:
- SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma): Smoldering multiple myeloma (SMM)is a premalignant plasma cell proliferative disorder. Multiple myeloma is a plasma cell neoplasm.
Arm/Group | MGUS (Monoclonal Gammopathy of Undetermined Significance) | SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma)
Number analyzed (Participants) | 10 | 17
pg/ml
  Ang2 (angiopoietin) | 2465.97 (589.27) | 3804.42 (467.16)
  G-CSF (granulocyte-colony stimulating factor) | 24.92 (11.66) | 101.08 (42.81)
  Follistatin | 562.45 (88.89) | 823.15 (83.00)
  HGF (hepatocyte growth factor) | 390.57 (70.82) | 654.34 (57.97)
  VEGF-A (vascular endothelial growth factor-A) | 844.31 (435.94) | 1301.52 (196.47)
  FGF-1 (fibroblast growth factor 1) | NA (NA) — Serum measures of FGF-1 were below the range of detectability, so these markers were excluded from analysis. | NA (NA) — Serum measures of FGF-1 were below the range of detectability, so these markers were excluded from analysis.
  Endothelin 1 | NA (NA) — Serum measures of endothelin-1 were below the range of detectability, so these markers were excluded from analysis. | NA (NA) — Serum measures of endothelin-1 were below the range of detectability, so these markers were excluded from analysis.
Statistical Analysis 1: Comparison: MGUS (Monoclonal Gammopathy of Undetermined Significance) vs SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma); Test type: Superiority; p = 0.024, Wilcoxon rank sum test — The reported p-value is representative of the difference in levels of Ang2 in both groups
Statistical Analysis 2: Comparison: MGUS (Monoclonal Gammopathy of Undetermined Significance) vs SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma); Test type: Superiority; p = 0.055, Wilcoxon rank sum test — The reported p-value is representative of the difference in levels of G-CSF in both groups
Statistical Analysis 3: Comparison: MGUS (Monoclonal Gammopathy of Undetermined Significance) vs SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma); Test type: Superiority; p = 0.055, Wilcoxon rank sum test — The reported p-value is representative of the difference in levels of Follistatin in both groups
Statistical Analysis 4: Comparison: MGUS (Monoclonal Gammopathy of Undetermined Significance) vs SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma); Test type: Superiority; p = 0.0098, Wilcoxon rank sum test — The reported p-value is representative of the difference in levels of HGF in both groups
Statistical Analysis 5: Comparison: MGUS (Monoclonal Gammopathy of Undetermined Significance) vs SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma); Test type: Superiority; p = 0.02, Wilcoxon rank sum test — The reported p-value is representative of the difference in levels of VEGF-A in both groups

4. Secondary Outcome: Comparison of Microvessel Density (MVD) Among Patients With MGUS, SMM, and MM
Description: Microvessel density was estimated by determining the average number of cluster of differentiation 34 (CD34)-stained microvessels in 10 areas of maximal MVD counted at a high-power field (h.p.f. x 500 magnification). Large vessels and vessels in the periosteum on bone were excluded. Areas of staining with no discrete breaks were counted as a single vessel. The presence of a lumen was not required.
Time Frame: 60 days
Population: Three patients with MM did not undergo bone marrow biopsies and were not included in this analysis.
Measure: Median (Full Range); unit: microvessels/hpf
Arm/Group | MGUS (Monoclonal Gammopathy of Undetermined Significance) | SMM (Smoldering Multiple Myeloma) | MM (Multiple Myeloma)
Number analyzed (Participants) | 10 | 10 | 7
microvessels/hpf | 15 [15 to 19.7] | 19.4 [7.6 to 32.5] | 20.9 [10.5 to 37.6]
Statistical Analysis 1: Comparison: MGUS (Monoclonal Gammopathy of Undetermined Significance) vs SMM (Smoldering Multiple Myeloma) vs MM (Multiple Myeloma); Test type: Other — Other, trend test; p = 0.008, Jonckheere-Terpstra test for trend

5. Secondary Outcome: Comparison of Reverse Contrast Transfer Rate (Kep) and Forward Contrast Transfer Rate (Ktrans) Among Patients With MGUS, SMM, and MM
Description: Pharmacokinetic parameters Kep and Ktrans were measured by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI).
Time Frame: 60 days
Population: Three patients with MM did not undergo bone marrow biopsies and were not included in this analysis.
Measure: Median (Full Range); unit: per min
Arm/Group | MGUS (Monoclonal Gammopathy of Undetermined Significance) | SMM (Smoldering Multiple Myeloma) | MM (Multiple Myeloma)
Number analyzed (Participants) | 10 | 10 | 7
per min
  Kep | 3.9 [1.6 to 9.2] | 9 [0.7 to 12.2] | 5.8 [2.1 to 12.7]
  Ktrans | 2.4 [1 to 4.2] | 2.3 [0.4 to 4.4] | 3.1 [1.6 to 4.1]
Statistical Analysis 1: Comparison: MGUS (Monoclonal Gammopathy of Undetermined Significance) vs SMM (Smoldering Multiple Myeloma) vs MM (Multiple Myeloma); Test type: Other — Other, trend test; p = 0.15, Jonckheere-Terpstra test for trend — The reported p-value is representative of the difference in levels of Kep between MGUS and SMM+MM
Statistical Analysis 2: Comparison: MGUS (Monoclonal Gammopathy of Undetermined Significance) vs SMM (Smoldering Multiple Myeloma) vs MM (Multiple Myeloma); Test type: Other — Other, trend test; p = 0.33, Jonckheere-Terpstra test for trend — The reported p-value is representative of the difference in levels of Ktrans between MGUS and SMM+MM

6. Secondary Outcome: Comparison of Serum Angiogenic Marker Reverse Contrast Transfer Rate (Kep) Between MGUS and SMM/MM Groups
Description: Pharmacokinetic parameter Kep was measured by dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI).
Time Frame: 60 days
Population: Serum was not available for three patients in the SMM group.
Measure: Mean (Standard Error); unit: per min
Arm/Group | MGUS (Monoclonal Gammopathy of Undetermined Significance) | SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma)
Number analyzed (Participants) | 10 | 17
per min | 4.05 (0.73) | 6.93 (0.97)
Statistical Analysis 1: Comparison: MGUS (Monoclonal Gammopathy of Undetermined Significance) vs SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma); Test type: Superiority; p = 0.08, Wilcoxon rank sum test

7. Secondary Outcome: Comparison of Microvessel Density (MVD) Between MGUS and SMM/MM Groups
Description: Microvessel density was estimated by determining the average number of CD34-stained microvessels in 10 areas of maximal MVD counted at a high-power field (h.p.f. x 500 magnification).
Time Frame: 60 days
Population: Serum was not available for three patients in the SMM group.
Measure: Mean (Standard Error); unit: microvessels/hpf
Arm/Group | MGUS (Monoclonal Gammopathy of Undetermined Significance) | SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma)
Number analyzed (Participants) | 10 | 17
microvessels/hpf | 15.04 (1.14) | 21.64 (1.90)
Statistical Analysis 1: Comparison: MGUS (Monoclonal Gammopathy of Undetermined Significance) vs SMM (Smoldering Multiple Myeloma)/MM (Multiple Myeloma); Test type: Superiority; p = 0.011, Wilcoxon rank sum test

ADVERSE EVENTS:
Arm/Group | Imaging in MGUS, SMM, and MM
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No